CLINICAL TRIAL: NCT04489628
Title: Tele-health Enabled Clinical Trial for COVID-19: Vitamin D as an Immunomodulator to Prevent Complications and Reduce Resource Utilization in Outpatients
Brief Title: Tele-health Enabled Clinical Trial for COVID-19
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to overcome hurdles to study recruitment
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Dr. Kevin Cooper, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20200461
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV Infection
Keywords: Vitamin D; Telehealth; SARS-CoV-2; Immune Storm
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Vitamin D (Active Comparator): Participants will be given 8 capsules of either cholecalciferol 50,000 IU or placebo at study randomization. Participants will be instructed to take 4 capsules on receipt of the treatment package(Day 0), 2 capsules on Day 5, 1 capsule on Day 10, and 1 capsule on Day 15. A phone or text reminder will be included at Days 5, 10, and 15 to take the additional doses of vitamin D.
  Interventions: Drug: Vitamin D3 or Placebo; Device: Doctella telehealth monitoring
- Placebo (Placebo Comparator): Participants will be given 8 capsules of either cholecalciferol 50,000 IU or placebo at study randomization. Participants will be instructed to take 4 capsules on receipt of the treatment package(Day 0), 2 capsules on Day 5, 1 capsule on Day 10, and 1 capsule on Day 15. A phone or text reminder will be included at Days 5, 10, and 15 to take the additional doses of vitamin D.
  Interventions: Device: Doctella telehealth monitoring

INTERVENTIONS:
Drug: Vitamin D3 or Placebo — ): Participants will be given 8 capsules of either cholecalciferol 50,000 IU or placebo at study randomization. Participants will be instructed to take 4 capsules on receipt of the treatment package(Day 0), 2 capsules on Day 5, 1 capsule on Day 10, and 1 capsule on Day 15. A phone or text reminder will be included at Days 5, 10, and 15 to take the additional doses of vitamin D.
  Arms: Vitamin D
Device: Doctella telehealth monitoring — Doctella device will be give to participants by the Emergency department as part of usual care to monitor heart rate, respiratory rate, oxygen saturation, and perfusion index vitals continuously for approximately 10 days. The study team will receive the vitals signs data (heart rate, respiratory rate, oxygen saturation, perfusion index, and temperature) retrospectively and will not be able to monitor patients in real time.

SUMMARY:
To determine the efficacy of high dose Vitamin D (an over-the-counter nutritional supplement) in preventing immune-related complications in outpatients with confirmed SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Laboratory confirmed SARS-CoV-2 infection < 4 days before randomization
3. Report of symptoms consistent with SARS-CoV-2 infection (including but not limited to fever, cough, muscle aches, joint pain, change in taste, change in smell, or shortness of breath) <4 days before admission
4. Asymptomatic or mild symptoms (not requiring hospital admission)
5. Access to and ability to use a mobile phone with telehealth capability

Exclusion Criteria:

1. Unable to provide informed consent or comply with study directions
2. Admitted to an acute care bed
3. Baseline serum calcium < 8.8 mg/dL or > 10.2 mg/dl (as evaluated by labs taken in the ER/urgent care)
4. Women who are currently breastfeeding
5. History of kidney stone in the past year or h/o multiple (>1) previous kidney stones
6. Does not have a smart phone that can download apps from Google Play or App Store.
7. No way to keep the phone charged consistently
8. The smartphone is shared with another individual.
9. Required laboratory data is unavailable (eg calcium levels)
10. No new oxygen requirement (see remote monitoring document)
11. Pregnant and lactating mothers.
12. Vitamin D level of 80ng/ml and above
13. No lab work for calcium or vitamin D completed in ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Patients requiring admission to the hospital or experiencing death | Days 1 to 15
  Proportion of patients requiring admission to the hospital or experiencing death by Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Wesley Yu, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No